CLINICAL TRIAL: NCT01910090
Title: Comparative, Randomized, Two-period, Two-treatment, Two-sequence, Single Dose, Open-label, Crossover Bioequivalence Study of FLURBIPROFEN 100 mg FAMOTIDINE 20 mg MULTI-LAYER TABLET (One Tablet) of (Sanovel İlaç San. ve Tic. A.Ş., İstanbul / Türkiye) Versus ANTADYS® Flurbiprofen 100 mg Comprimé Pelliculé (One Film-coated Tablet) of (LaboratoireThẻramex 6, Avenue Albert II- BP.59 98007 MONACO Cedex) and PEPCID® (Famotidine) 20 mg Tablets, USP (One Tablet) of (Marathon Pharmaceuticals, LLC USA) in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of FLURBIPROFEN 100 mg FAMOTIDINE 20 mg MULTI-LAYER TABLET in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Research Unit, Jordan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: FAFL439/PRO-00
Record Dates: First submitted 2012-12-15; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: fasting condition
MeSH Terms: interventions — Flurbiprofen; Famotidine

ARMS (2):
- FLURBIPROFEN 100 mg FAMOTIDINE 20 mg MULTI-LAYER TABLET (Experimental): FLURBIPROFEN, FAMOTIDINE 100/20 mg MULTI-LAYER TABLET one tablet, once
  Interventions: Drug: FLURBIPROFEN 100 mg FAMOTIDINE 20 mg MULTI-LAYER TABLET
- ANTADYS® and PEPCID® (Active Comparator): ANTADYS® 100 mg, PEPCID® 20 mg two tablets, taken once
  Interventions: Drug: ANTADYS® 100 mg, PEPCID® 20 mg

INTERVENTIONS:
Drug: FLURBIPROFEN 100 mg FAMOTIDINE 20 mg MULTI-LAYER TABLET — MULTI-LAYER TABLET
  Other Names: MULTI-LAYER TABLET
  Arms: FLURBIPROFEN 100 mg FAMOTIDINE 20 mg MULTI-LAYER TABLET
Drug: ANTADYS® 100 mg, PEPCID® 20 mg — ANTADYS® 100 mg, PEPCID® 20 mg two tablets, taken once
  Other Names: ANTADYS® 100 mg, PEPCID® 20 mg two tablets, taken once
  Arms: ANTADYS® and PEPCID®

SUMMARY:
To assess the bioequivalence of Test oral formulation of FLURBIPROFEN 100 mg FAMOTIDINE 20 mg MULTI-LAYER TABLET versus Reference ANTADYS®100 mg Comprimé Pelliculé & PEPCID® (Famotidine) 20mg Tablets, USP.

DETAILED DESCRIPTION:
An open-label, randomized, single dose, two-treatment, two-period, two-sequence, crossover bioequivalence with a washout period of at least 7 days between doses Healthy mixed skin Arab & Mediterranean Subjects ages between 18 and 45 years, body-mass index 18.5 to 30.0 kg/m2 inclusive, non-smokers or light smokers (smokers of not more than 10 cigarettes per day).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male subjects.
2. Ethnic Group: Arab & Mediterranean
3. Race: Mixed skin (white & black skin people).
4. Age 18-45 years
5. Body-mass index 18.5 to 30.0 kg/m2 inclusive
6. Subject is available for the whole study period and gave written informed consent
7. Physical examination within normal ranges
8. All laboratory screening results within the normal range, or being assessed as clinically non-significant by the attending physician.
9. Vital signs within normal ranges (Unless clinical investigator classified as insignificant).
10. Normal Kidney & Liver function tests (Unless clinical investigator classified as insignificant).
11. Normal Cardiovascular system.
12. Normal Digestive system.

Exclusion Criteria:

1. Women.
2. Ethnic Group (Non- Arab &/ or Non- Mediterranean)
3. History of severe allergy or allergic reactions to study drug or related drugs
4. Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
5. History of serious illness that can impact fate of drugs
6. Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, unless judged not clinically significant by the Principal Investigator, or medical designate
7. Clinically significant illness 4 weeks before study Period I
8. Mental disease, drug, alcohol, solvents or caffeine abuse, smoking.
9. Regular use of medication
10. Having taken medication that could affect the investigated drug product: a) Regular consumption of drugs during the two weeks prior to study initiation day, b) consumption of enzyme stimulating or inhibiting drugs (e.g. Barbiturates, Carbamazepine, Phenytoin) during one month before the study initiation.
11. Presence of any significant physical or organ abnormality
12. Donation of 1) at least 400 ml of blood within 60 days, or 2) more than 150 ml of blood within 30 days, or 3) more than 100 ml blood plasma or platelets within 14 days before study Period I
13. Participation in another bioequivalence study within 80 days prior to the start of this study Period I
14. Following a special diet (e.g. vegetarian) or dieting one month before the study initiation.
15. History of Gastrointestinal diseases
16. Prior history of hypersensitivity to Flurbiprofen or Famotidine and other competitive inhibitor of histamine H2-receptors.
17. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration
18. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
19. Exhausting physical exercise in the last 48 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
20. Any significant clinical abnormality including HBsAg, HCV, and HIV
21. Abnormal vital signs
22. Abnormal Kidney or Liver function tests.
23. Abnormal Cardiovascular system.
24. Abnormal Digestive system
25. Vomiting, Diarrhea.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
cmax | five weeks
  Cmax Ratio: The 90% confidence interval for this measure lies within an acceptance range of 80.00% - 125.00% based on Flurbiprofen and Famotidine.
  AUC Ratio: The 90% confidence interval for this measure lies within an acceptance range of 80.00% - 125.00% based on Flurbiprofen and Famotidine.
tmax | three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rana T. Bustami, Ph.D. of Pharmacy, Principal Investigator — PRU; Dr. Rana T. Bustami, Ph.D. of Pharmacy, Principal Investigator — Dr. Rana T. Bustami
Locations (1):
- Arab Pharmaceutical industry Consulting/ Pharmaceutical Research Unit, Amman, Jordan